CLINICAL TRIAL: NCT00709826
Title: APRiCOT-P (Apricoxib in Combination Oncology Treatment - Pancreas): Phase 2 Study of the Efficacy and Safety of Apricoxib in Combination With Gemcitabine and Erlotinib in the Treatment of Patients With Advanced Pancreatic Cancer
Brief Title: APRiCOT-P: Study of Apricoxib With Gemcitabine and Erlotinib to Treat Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tragara Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TP2001-203; APRiCOT-P (Other: Tragara Pharmaceuticals)
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Results first posted 2012-11-07 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-10

CONDITIONS: Pancreatic Cancer; Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Erlotinib Hydrochloride; apricoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- apricoxib + gemcitabine + erlotinib (Experimental): 400mg apricoxib + 1000mg/m2 gemcitabine + 100mg erlotinib
  Interventions: Drug: gemcitabine; Drug: Erlotinib; Drug: apricoxib
- placebo + gemcitabine + erlotinib (Placebo Comparator): placebo + 1000mg/m2 gemcitabine + 100mg erlotinib
  Interventions: Drug: gemcitabine; Drug: placebo; Drug: Erlotinib

INTERVENTIONS:
Drug: gemcitabine — Gemcitabine: per package insert.
  Other Names: Gemcitabine - Gemzar
Drug: placebo — placebo: 100 mg tablets, 400 mg/day
  Other Names: No other names
  Arms: placebo + gemcitabine + erlotinib
Drug: Erlotinib — Erlotinib - per package insert.
  Other Names: Erlotinib - Tarceva
Drug: apricoxib — apricoxib: 100mg tablets, given orally
  Other Names: No other names
  Arms: apricoxib + gemcitabine + erlotinib

SUMMARY:
This study will compare the anti-tumor efficacy of apricoxib and gemcitabine/erlotinib with placebo and gemcitabine/erlotinib in patients with advanced pancreatic cancer.

DETAILED DESCRIPTION:
This study will compare the anti-tumor efficacy of apricoxib and gemcitabine/erlotinib with placebo and gemcitabine/erlotinib as measured by progression-free survival to test the hypothesis that down regulation of COX-2 and EGFR pathways in patients with up-regulated COX-2 expression in tumors will have a clinical benefit compared with Gemcitabine/Erlotinib only.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed adenocarcinoma of the pancreas that is locally advanced or metastatic.
2. Life expectancy greater than or equal to 3 months.
3. Patients must have measurable disease by RECIST.
4. ECOG PS of 0, 1, or 2.
5. Negative serum pregnancy test at the time of first dose for women of childbearing potential.

Exclusion Criteria:

1. Previous chemotherapy as primary treatment for locally advanced or metastatic pancreatic cancer(stage 3 T3 and T4, and all stage 4).
2. RT within 2 weeks or chemotherapy within 3 weeks or noncytotoxic investigational agents within 4 weeks of initiating study treatment.
3. Evidence of New York Heart Association class III or greater cardiac disease.
4. History of myocardial infarction, stroke, ventricular arrhythmia.
5. Symptomatic central nervous system metastases.
6. Pregnant or nursing women.
7. Hypersensitivity or intolerance to apricoxib, erlotinib, gemcitabine, sulfonamides, aspirin, or other non-steroidal anti-inflammatory drugs (NSAIDs).
8. History of upper gastrointestinal bleeding, ulceration or perforation. History of lower GI bleeding, ulceration, or perforation within 12 months.
9. Previous anti-EGFR kinase therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2008-08; Primary Completion 2010-06 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Parrott, Study Director — Tragara Pharmaceuticals, Inc.
Locations (39):
- United States (39):
  - Arizona Clinical Research Center, Tucson, Arizona
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - Southbay Oncology Hematology Partners, Campbell, California
  - Bay Area Cancer Research Group, LLC, Concord, California
  - Bay Area Cancer Research Group, LLC, Pleasant Hill, California
  - North America Research Institute, San Dimas, California
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Oncology Associates of Bridgeport, Trumball, Connecticut
  - Hematology Oncology Associates, Lake Worth, Florida
  - Hematology Oncology Associates of Treasure Coast, Port Saint Lucie, Florida
  - The Queen's Medical Center Cancer Center, Honolulu, Hawaii
  - Rush-Copley Medical Center, Aurora, Illinois
  - Alexian Brothers Medical Hospital Network, Elk Grove Village, Illinois
  - Investigative Clinical Research of Indiana, LLC, Indianapolis, Indiana
  - Medical Consultants, PC, Muncie, Indiana
  - University of Iowa Hospitals, Iowa City, Iowa
  - Owsley Brown Frazier Cancer Center, Louisville, Kentucky
  - Jayne Gurtler, MD, Metairie, Louisiana
  - Franklin Square Hospital Center/Harry and Jeanette Weinberg Cancer Institute at Franklin Square, Baltimore, Maryland
  - SJMH Cancer Center, Ann Arbor, Michigan
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Warren Hospital, Phillipsburg, New Jersey
  - San Juan Oncology Associates, Farmington, New Mexico
  - Bronx River Medical Associates, P.C., The Bronx, New York
  - Cancer Care of WNC, PA, Asheville, North Carolina
  - Southeastern Medical Oncology Center, Goldsboro, North Carolina
  - Southeastern Medical Oncology Center, Wilson, North Carolina
  - Samaritan Hematology * Oncology, Corvallis, Oregon
  - Eastern Regional Medical Center, Philadelphia, Pennsylvania
  - Associates in Hematology-Oncology PC, Upland, Pennsylvania
  - Berks Hematology-Oncology Associates, Ltd, West Reading, Pennsylvania
  - Charleston Hematology Oncology Associates, Charleston, South Carolina
  - JTV Cancer Care Institute, Rapid City, South Dakota
  - The Jones Clinic, Germantown, Tennessee
  - Tennessee Cancer Specialists, Knoxville, Tennessee
  - Coastal Bend Cancer Center, Corpus Christi, Texas
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - The Methodist Hospital, Houston, Texas
  - Cascade Cancer Center, Kirkland, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study opened to accrual in August 2008. Enrollment closed on November 2010. One hundred and nine patients were randomized. Patients were recruited from clinical oncology practices.
Groups:
- Apricoxib/Gemcitabine/Erlotinib: Patients randomized to receive apricoxib + gemcitabine + erlotinib.
- Placebo/Gemcitabine/Erlotinib: Patients randomized to receive placebo + gemcitabine + erlotinib.
Period: Overall Study
Arm/Group | Apricoxib/Gemcitabine/Erlotinib | Placebo/Gemcitabine/Erlotinib
Started | 70 | 39
Completed | 68 | 38
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Apricoxib/Gemcitabine/Erlotinib | Placebo/Gemcitabine/Erlotinib | Total
Number analyzed (Participants) | 70 | 39 | 109
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 17 | 55
  >=65 years | 32 | 22 | 54
Age Continuous [Mean (Standard Deviation); unit: years] | 63 (64.2) | 67 (66) | 64 (64.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 22 | 63
  Male | 29 | 17 | 46
Region of Enrollment [Number; unit: participants]
  United States | 70 | 39 | 109

OUTCOME MEASURES:

1. Secondary Outcome: Overall Survival
Time Frame: Randomization then every other cycle
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Apricoxib/Gemcitabine/Erlotinib | Placebo/Gemcitabine/Erlotinib
Number analyzed (Participants) | 70 | 39
Months | 5.0 [3.67 to 50.47] | 4.8 [4.07 to 5.70]

2. Primary Outcome: Progression Free Survival
Description: Progression is defined, using RECIST, as a measurable increase in the smallest dimension of any target or non-target lesion, or the appearance of new lesions, since baseline.
Time Frame: Randomization then every other cycle
Population: A 1-sided log rank test was used to achieve 80% power at an α=0.20 significance level to detect a difference of 0.16 between the proportions of patients who were progression free in AP/EG (0.35) and P/EG (0.19) after 9 months; an overall sample size of approximately 110 patients (73 in AP/EG and 37 in P/EG) was randomized in a 2:1 ratio.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Apricoxib/Gemcitabine/Erlotinib | Placebo/Gemcitabine/Erlotinib
Number analyzed (Participants) | 70 | 39
Months | 3.0 [2.57 to 6.47] | 2.8 [2.63 to 4.60]

ADVERSE EVENTS:
Time Frame: First dose of study drug to 30 days after last dose of study drug
Description: Only drug-related serious adverse events are listed.
Arm/Group | Apricoxib/Gemcitabine/Erlotinib | Placebo/Gemcitabine/Erlotinib
Serious Adverse Events (participants affected / at risk) | 16/70 | 5/39
Other Adverse Events (participants affected / at risk) | 70/70 | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apricoxib/Gemcitabine/Erlotinib (N=70) | Placebo/Gemcitabine/Erlotinib (N=39)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 5 (5) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophagitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
International normalized ratio increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Vascular disorders) | 1 (1) | 0 (0)
Embolic stroke (Vascular disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apricoxib/Gemcitabine/Erlotinib (N=70) | Placebo/Gemcitabine/Erlotinib (N=39)
Diarrhea (Gastrointestinal disorders) | 41 (41) | 17 (17)
Nausea (Gastrointestinal disorders) | 41 (41) | 15 (15)
Fatigue (General disorders) | 40 (40) | 24 (24)
Anemia (Blood and lymphatic system disorders) | 37 (37) | 18 (18)
Rash (Skin and subcutaneous tissue disorders) | 32 (32) | 20 (20)
Thrombocytopenia (Blood and lymphatic system disorders) | 29 (29) | 14 (14)
Constipation (Gastrointestinal disorders) | 26 (26) | 7 (7)
Vomiting (Gastrointestinal disorders) | 23 (23) | 12 (12)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 22 (22) | 14 (14)
Abdominal pain (Gastrointestinal disorders) | 21 (21) | 6 (6)
Neutropenia (Blood and lymphatic system disorders) | 21 (21) | 13 (13)
Edema peripheral (Musculoskeletal and connective tissue disorders) | 21 (21) | 18 (18)
Anorexia (Metabolism and nutrition disorders) | 18 (18) | 6 (6)
Dehydration (General disorders) | 17 (17) | 6 (6)
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 15 (15) | 2 (2)
Mucosal inflammation (Gastrointestinal disorders) | 12 (12) | 4 (4)
Insomnia (Psychiatric disorders) | 11 (11) | 5 (5)
Abdominal distension (Gastrointestinal disorders) | 10 (10) | 3 (3)
Dizziness (Nervous system disorders) | 10 (10) | 5 (5)
Hypokalemia (Metabolism and nutrition disorders) | 10 (10) | 6 (6)
Asthenia (General disorders) | 9 (9) | 6 (6)
Dyspepsia (Gastrointestinal disorders) | 9 (9) | 1 (1)
Chills (General disorders) | 8 (8) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 5 (5)
Deep vein thrombosis (Vascular disorders) | 8 (8) | 5 (5)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 8 (8) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 7 (7) | 3 (3)
Anxiety (Psychiatric disorders) | 7 (7) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 3 (3)
Epistaxis (Vascular disorders) | 7 (7) | 4 (4)
Hypotension (Vascular disorders) | 7 (7) | 5 (5)
Night sweats (Skin and subcutaneous tissue disorders) | 7 (7) | 1 (1)
Ascites (Gastrointestinal disorders) | 6 (6) | 1 (1)
Flatulence (Gastrointestinal disorders) | 6 (6) | 0 (0)
Jaundice (Hepatobiliary disorders) | 6 (6) | 3 (3)
Pneumonia (Infections and infestations) | 6 (6) | 2 (2)
Renal failure (Renal and urinary disorders) | 6 (6) | 0 (0)
Weight decreased (Investigations) | 6 (6) | 4 (4)
Alanine aminotransferase increased (Investigations) | 5 (5) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (4)
Cellulitis (Infections and infestations) | 5 (5) | 1 (1)
Depression (Psychiatric disorders) | 5 (5) | 5 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2)
Dysgeusia (Nervous system disorders) | 5 (5) | 4 (4)
Headache (Nervous system disorders) | 5 (5) | 2 (2)
Liver function test abnormal (Investigations) | 5 (5) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 6 (6)
Pyrexia (General disorders) | 5 (5) | 7 (7)
Stomatitis (Gastrointestinal disorders) | 5 (5) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 5 (5)
Erythema (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 2 (2)
Hyperbilirubinemia (Hepatobiliary disorders) | 4 (4) | 3 (3)
Edema (General disorders) | 4 (4) | 2 (2)
Pain (General disorders) | 4 (4) | 3 (3)
Pulmonary embolism (Vascular disorders) | 4 (4) | 4 (4)
Urinary tract infection (Infections and infestations) | 4 (4) | 7 (7)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2) | 6 (6)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No